CLINICAL TRIAL: NCT00614913
Title: Phase I/II Study of Proton Beam Therapy for Hepatocellular Carcinoma
Brief Title: Proton Beam Therapy for Treatment of Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, David Bush, Principal Inverstigator, Loma Linda University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSR #48095
Record Dates: First submitted 2007-12-26; First posted 2008-02-13 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-07

CONDITIONS: Liver Cancer; Hepatocellular Carcinoma
Keywords: Proton; Radiotherapy; Hepatocellular carcinoma; Liver Cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Proton radiation therapy — A total dose of 63 Gy will be delivered in 15 equally divided daily fractions over a 3 week coarse as an out-patient.

SUMMARY:
This study is designed to evaluate the possible benefits and side effects of the use of proton therapy for patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a type of primary cancer of the liver that is being diagnosed in the U.S. population with increasing frequency. While surgery is the first line of treatment, many patients are not eligible for surgical removal. Current non-surgical treatments for HCC are not fully effective and can have substantial side-effects. This study utilizes a type of radiation treatment called proton beam that can deliver high doses of radiotherapy to tumors within the liver while minimizing damage to surrounding healthy tissues. The treatment is non-invasive and is given on an out-patient basis over a three week coarse. The study will evaluate the effectiveness and side-effects of this therapy by tracking patient's outcomes following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hepatocellular carcinoma
* Adult patients aged 18 years old and above
* Ability to give informed consent for study
* Compensated liver disease

Exclusion Criteria:

* Pediatric patients (aged less than 18 years old)
* Decompensated or advanced liver disease
* Poorly controlled ascites
* Variceal hemorrhage within the previous 30 days
* Recurrent hepatic encephalopathy
* Cirrhosis with CTP* score >10
* Active alcohol or drug abuse
* Anticipated survival of less than 30 days
* Advanced co-morbid medical illnesses
* Karnofsky Performance Score <60

Tumor characteristics:

- Any tumor that can not be safely and effectively irradiated due to inability to deliver target treatment dose to required treatment volume or due to prohibitively high risk of anticipated toxicities to normal liver or nearby bowel, stomach, kidney or spinal cord.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 1998-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Bush, MD, Principal Investigator — Loma Linda University Dept. of Radiation Medicine; Jerry D Slater, MD, Study Chair — Loma Linda University Department of Radiation Medicine
Locations (1):
- Loma Linda University Medical Center / James M. Slater Proton Treatment Center, Loma Linda, California, United States

REFERENCES:
- [Result] Bush DA, Hillebrand DJ, Slater JM, Slater JD. High-dose proton beam radiotherapy of hepatocellular carcinoma: preliminary results of a phase II trial. Gastroenterology. 2004 Nov;127(5 Suppl 1):S189-93. doi: 10.1053/j.gastro.2004.09.033. PMID 15508084
- [Result] Bush DA, Kayali Z, Grove R, Slater JD. The safety and efficacy of high-dose proton beam radiotherapy for hepatocellular carcinoma: a phase 2 prospective trial. Cancer. 2011 Jul 1;117(13):3053-9. doi: 10.1002/cncr.25809. Epub 2011 Jan 24. PMID 21264826

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with a diagnosis of hepatocellular carcinoma were recruited from the hepatology clinic at Loma Linda University Medical Center to participate in this trial.
Pre-assignment Details: Patients with documented metastatic disease were excluded from this trial.
Groups:
- Proton Beam Therapy: Patients received 63Gy in three weeks with proton beam.
Period: Overall Study
Arm/Group | Proton Beam Therapy
Started | 76
Completed | 76
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Proton Beam Therapy
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 62.7 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 53
Region of Enrollment [Number; unit: participants]
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: 3-year Survival Without Tumor Progression for Patients Within the Milan Criteria
Description: Percent of participants alive and without tumor progression 3 years following treatment.
Time Frame: 3 months
Population: Participants that were within the Milan criteria
Measure: Number; unit: percentage of participants
Arm/Group | Proton Beam Therapy
Number analyzed (Participants) | 35
percentage of participants | 60

2. Primary Outcome: Median Survival Without Tumor Progression
Description: Median time until disease progression or death
Time Frame: 3 months
Population: All participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Proton Beam Therapy
Number analyzed (Participants) | 76
months | 36 [16 to 56]

ADVERSE EVENTS:
Arm/Group | Proton Beam Therapy
Serious Adverse Events (participants affected / at risk) | 5/76
Other Adverse Events (participants affected / at risk) | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Beam Therapy (N=76)
GI Bleeding (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes